CLINICAL TRIAL: NCT02244164
Title: Pathophysiological Study of the Increase in Pancreatic Volume in Type 2 Diabetes Treatments.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too slow
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Incretine study
Record Dates: First submitted 2014-09-15; First posted 2014-09-18 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes; Incretinomimetics; Pancreas
Keywords: Type 2 Diabetes; Incretinomimetics; DPP-4 inhibitors; Pancreas; PanIN; RMN; Lipasemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Liraglutide; lixisenatide; Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate; Vildagliptin; saxagliptin; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sulfonylurea (Active Comparator): Patient will received metformine with sulfonylurea
  Interventions: Drug: Incretinomimetics; Drug: DPP-4 inhibitors
- Incretinomimectics (Active Comparator): Patients will received metformin with sulfonylurea with GLP-1 analogue
  Interventions: Drug: DPP-4 inhibitors
- DPP-4 inhibitors (Active Comparator): Patients will received metformin with DPP-4 inhibitors
  Interventions: Drug: Incretinomimetics

INTERVENTIONS:
Drug: Incretinomimetics
  Other Names: - exenatide (Byetta®); - liraglutide (Victoza®); - lixisenatide (Lyxumia®); - exenatide extended-release (Bydureon®).
  Arms: DPP-4 inhibitors; Sulfonylurea
Drug: DPP-4 inhibitors
  Other Names: - sitagliptine (Januvia®); - vildagliptine (Galvus®); - saxagliptine (Onglyza®); - linagliptine (Trajenta®).
  Arms: Incretinomimectics; Sulfonylurea

SUMMARY:
Incretinomimetics and inhibitors of dipeptidyl peptidase-4 (DPP-4) are new treatments for diabetes. Previous retrospective studies have shown that these treatments induced an increase in pancreatic mass with potentially a risk for pancreatitis and development of precancerous lesions.

The aim of our study is to provide a better understanding of the pathophysiological mechanisms of increased volume and / or pancreatic exocrine secretion when exposed to certain treatment of type 2 diabetes.

DETAILED DESCRIPTION:
The incretinomimetics and the inhibitors of dipeptidyl peptidase-4 (DPP-4) are new treatments for diabetes. The incretinomimetics are analogs of Glucagon Like Peptide 1 (GLP-1), secreted from endocrine L-cells of the colon and terminal ileum peptide. Serum GLP-1 increase rapidly after a meal. But its degradation is also fast. It acts on the hypothalamus by reducing appetite and food intake, on the stomach by delaying gastric emptying and the level of beta islet cells by inducing the synthesis and secretion of insulin (1). The incretinomimetics currently marketed in Belgium (March 2014) are exenatide (Byetta ®), liraglutide (Victoza ®), lixisenatide (Lyxumia ®) and very soon (April 2014) extended-release exenatide (Bydureon ®). The DPP-4 prevent the degradation of GLP-1. The DPP-4 currently marketed (March 2014) are sitagliptin (Januvia ®), vildagliptin (Galvus ®), saxagliptin (Onglyza ®) and (Trajenta ®) linagliptin.

In diabetic patients, these treatments allow a significant reduction in fasting plasma glucose and postprandial, with a low risk of hypoglycemia and no weight gain (and sometimes weight loss) (2).

Their place in the management of type 2 diabetes is considered or in combination with metformin, when diabetes is inadequately controlled despite maximal dose of the latter, or when patients are intolerant to metformin.

A study to evaluate the safety of 'incretinomimetics therapy "showed an increase in pancreatic weight of 40% (3). Indeed, in a cohort of 34 pancreatic organ donors from brain death, 20 patients were diabetic and 8 as incretin mimetics for over 1 year. An increase in pancreatic mass on average 40% was observed compared to diabetic patients without this treatment.

This study also demonstrated an increase in the mass of beta cells without restoring insulin function. The advanced for this mass increase without a significant increase of cell size is a hypothesis decreased apoptosis of beta cells.

Furthermore there is also an increase in the mass of cells producing α intraductulaire cell proliferation. This would be responsible for the onset of pancreatitis but also the appearance of endocrine microadenomas. The same study (3) also observed an increase in cell proliferation in the exocrine compartment of the pancreas (ductal and acinar cells) induced by incretinomimetic and an increased frequency of lesions potentially pre-cancerous PanIN 1 and 2 with this treatment.

Another study (4) by the same group of researchers showed that GLP-1 induced ductal cell growth in rats treated with high-dose exenatide for 12 weeks. It could therefore, by ductal obstruction induce pancreatitis.

All of these studies therefore warns about these new treatments potentially inducers of different pancreatic lesions.

The aim of our study is to provide a better understanding of the pathophysiological mechanisms of increased volume and / or pancreatic exocrine secretion when exposed to certain treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes inadequately controlled or intolerant to metformin
* Obtaining informed consent
* Aged between 18 and 70 years
* BMI between 20 and 45 kg / m²

Exclusion Criteria:

* Contraindication to nuclear magnetic resonance (NMR):
* Carrying a metallic foreign body (pacemaker, valve, intraocular equipment, clips)
* Allergy to Gadolinium / Secretin
* Pregnancy or breastfeeding
* Contraindication to treatment with incretinomimetic:
* Hypersensitivity to the active substance or to any of the excipients
* Severe Gastroparesis
* Severe renal impairment
* History of Surgery (gastroduodenal, pancreatic or ileocecal)
* Presence or history of pancreatic disease
* Active alcoholism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-10; Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Volumetric measurement of the pancreas | 1 year
  A RMN will be done before and 1 year after the treatment. A comparative mesure of pancreatic volume will be performed.

SECONDARY OUTCOMES:
Quantitative response to secretin | 1 year
  A RMN with injection of secretin will be done before and after the treatment. A quantitative evaluation of secretin response will be performed.

OTHER OUTCOMES:
Fasting glycemia | 1 year
  Quarterly during 1 years a blood analysis will be done.
C-Peptide | 1 years
  Quarterly during 1 year a blood analysis will be done.
HbA1c | 1 year
  Quarterly during 1 year a blood analysis will be done.
Cholesterol | 1 year
  Quarterly during 1 year a blood analysis will be done.
Calcium | 1 year
  Quarterly during 1 year a blood analysis will be done.
Phosphorus | 1 year
  Quarterly during 1 year a blood analysis will be done.
Urea | 1 year
  Quarterly during 1 year a blood analysis will be done.
Creatininemia | 1 year
  Quarterly during 1 year a blood analysis will be done.
Bilirubinemia | 1 year
  Quarterly during 1 year a blood analysis will be done.
Alcaline phosphatase | 1 year
  Quarterly during 1 year a blood analysis will be done.
Gamma GT | 1 year
  Quarterly during 1 year a blood analysis will be done.
Alanine aminotransferase | 1 year
  Quarterly during 1 year a blood analysis will be done.
Asparate aminotransferase | 1 year
  Quarterly during 1 year a blood analysis will be done.
Lipasemia | 1 year
  Quarterly during 1 year a blood analysis will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Huberty, MD, Principal Investigator — Gastroenterology Department Erasme Hospital
Locations (1):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium

REFERENCES:
- [Result] Drucker DJ, Nauck MA. The incretin system: glucagon-like peptide-1 receptor agonists and dipeptidyl peptidase-4 inhibitors in type 2 diabetes. Lancet. 2006 Nov 11;368(9548):1696-705. doi: 10.1016/S0140-6736(06)69705-5. PMID 17098089
- [Result] Amori RE, Lau J, Pittas AG. Efficacy and safety of incretin therapy in type 2 diabetes: systematic review and meta-analysis. JAMA. 2007 Jul 11;298(2):194-206. doi: 10.1001/jama.298.2.194. PMID 17622601
- [Result] Butler AE, Campbell-Thompson M, Gurlo T, Dawson DW, Atkinson M, Butler PC. Marked expansion of exocrine and endocrine pancreas with incretin therapy in humans with increased exocrine pancreas dysplasia and the potential for glucagon-producing neuroendocrine tumors. Diabetes. 2013 Jul;62(7):2595-604. doi: 10.2337/db12-1686. Epub 2013 Mar 22. PMID 23524641
- [Result] Butler PC, Elashoff M, Elashoff R, Gale EA. A critical analysis of the clinical use of incretin-based therapies: Are the GLP-1 therapies safe? Diabetes Care. 2013 Jul;36(7):2118-25. doi: 10.2337/dc12-2713. Epub 2013 May 3. PMID 23645885